CLINICAL TRIAL: NCT00537979
Title: Prospective, Non-randomized, Multicenter Study to Assess the Efficacy and Safety of Oral or Intravenous Paricalcitol Administered Over 6 Months to Patients With Secondary Hyperparathyroidism on Dialysis
Brief Title: Efficacy and Safety of 6 Months Treatment With Paricalcitol Injection or Oral in Patients With Secondary Hyperparathyroidism on Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W10-129
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-09

CONDITIONS: Secondary Hyperparathyroidism; Dialysis
Keywords: Dialysis; Hyperparathyroidism; Zemplar
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hyperparathyroidism | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol injection (Active Comparator): ABT-358 Zemplar
  Interventions: Drug: Paricalcitol injection
- Paricalcitol capsules (Active Comparator): ABT-358 Zemplar
  Interventions: Drug: Paricalcitol capsules

INTERVENTIONS:
Drug: Paricalcitol injection — Most recent iPTH level in pg/mL divided by 100 = dose in mcg; dose is rounded down to nearest mcg and administered 3x weekly
  Other Names: ABT-358; paricalcitol; Zemplar
  Arms: Paricalcitol injection
Drug: Paricalcitol capsules — Most recent iPTH level in pg/mL divided by 80 = dose in mcg; dose is rounded down to nearest mcg and administered 3x weekly
  Other Names: ABT-358; paricalcitol; Zemplar
  Arms: Paricalcitol capsules

SUMMARY:
Prospective, non-randomized, multi-center study to assess the efficacy and safety of paricalcitol injection or oral administered over 6 months to patients with secondary hyperparathyroidism on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years with secondary hyperparathyroidism (iPTH >= 300 pg/mL)
* Patients in a chronic hemodialysis or peritoneal dialysis program previously treated with vitamin D metabolites or without previous treatment
* Patients in which treatment with paricalcitol injection or oral is clinically indicated according to the criteria of the participating investigator
* Patients providing their signed informed consent to participate in the trial

Exclusion Criteria:

* Patients with severe hyperparathyroidism (iPTH > 3,000 pg/ml)
* Patients with hypercalcaemia (calcium >=11.0 mg/dl, adjusted according to Albumin level), hyperphosphataemia (phosphorus >= 6.5 mg/dl) or patients with calcium x phosphorus >= 70
* Known hypersensitivity and/or toxicity to vitamin D metabolites and/or other product ingredients
* Patients who have participated in clinical studies within the last month or who are currently enrolled in clinical studies
* Patients who cannot tolerate or take phosphorus binders that do not contain Calcium and/or Aluminum
* Patients that in the opinion of the investigator, for any reason, are not good candidates for therapy with Synthetic Analogues of Vitamin D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Luis Cañadas, MD, Study Director — Abbott
Locations (12):
- Mexico (12):
  - Site Ref # / Investigator 19391, Jojutla Morelos
  - Site Ref # / Investigator 19392, Mexico City
  - Site Ref # / Investigator 19397, Mexico City
  - Site Ref # / Investigator 19396, Mexico City
  - Site Ref # / Investigator 19389, Mexico City
  - Site Ref # / Investigator 19390, Mexico City
  - Site Ref # / Investigator 19393, Mexico City
  - Site Ref # / Investigator 19394, Mexico City
  - Site Ref # / Investigator 19395, Mexico City
  - Site Ref # / Investigator 19399, Puebla City
  - Site Ref # / Investigator 19398, Zapopan
  - Site Ref # / Investigator 19388, Zapopan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into the study at 12 dialysis centers in Mexico. Recruitment began in September 2007 and ended in January 2010. The study population consisted of patients on hemodialysis or peritoneal dialysis with a diagnosis of secondary hyperparathyroidism.
Groups:
- Paricalcitol Injection: Paricalcitol (ABT-358 Zemplar) Injection was administered to participants on hemodialysis.
- Paricalcitol Capsules: Paricalcitol (ABT-358 Zemplar) capsules were administered to participants on peritoneal dialysis.
Period: Overall Study
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules
Started | 38 | 109
Completed | 32 | 89
Not Completed | 6 | 20
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Non-compliance with treatment/procedure | 2 | 2
Not completed — Death | 0 | 3
Not completed — Kidney transplant | 0 | 3
Not completed — Heart failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules | Total
Number analyzed (Participants) | 38 | 109 | 147
Age Continuous [Mean (Standard Deviation); unit: years] | 43.79 (16.36) | 44.89 (17.91) | 44.39 (17.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 50 | 71
  Male | 17 | 59 | 76
Region of Enrollment [Number; unit: participants]
  Mexico | 38 | 109 | 147

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve at Least a 50% Reduction in iPTH Compared to Baseline Level
Description: Number of participants who achieved at least a 50% reduction in intact parathyroid hormone (iPTH) compared to the baseline level.
Time Frame: 24 weeks
Population: The analysis was intention to treat (ITT). The ITT population was defined as all participants who fulfilled inclusion criteria and received at least one dose of paricalcitol.
Measure: Number; unit: participants
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules
Number analyzed (Participants) | 38 | 109
participants | 17 | 57

2. Secondary Outcome: Analysis of Episodes of Hypercalcemia (> 11.5 mg/dL), Hyperphosphatemia (> 7.0 mg/dL) and Elevations of Calcium x Phosphorus Product (> 75)
Description: Number of participants with hypercalcemia (calcium levels greater than 11.5 mg/dL), hyperphosphatemia (phosphorus levels greater than 7.0 mg/dL), or calcium x phosphorus product levels greater than 75.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules
Number analyzed (Participants) | 38 | 109
participants
  Hypercalcemia | 2 | 6
  Hyperphosphatemia | 9 | 19
  Elevated calcium x phosphorus product | 3 | 14

3. Secondary Outcome: Proportion of Subjects Who Achieve an iPTH <300 pg/mL
Description: Number of participants who achieved an intact parathyroid hormone (iPTH) level of less than 300 pg/mL.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules
Number analyzed (Participants) | 38 | 109
participants | 16 | 57

4. Secondary Outcome: Time Required to Achieve: (1) a Reduction in iPTH Less Than <300 pg/mL;(2) a 50% Reduction in iPTH Compared to the Baseline Level; and (3) Either a Reduction in iPTH Less Than <300 pg/mL or a 50% Reduction in iPTH Compared to the Baseline Level
Description: Number of days required to achieve a reduction in intact parathyroid hormone (iPTH) to less than 300 pg/mL, a reduction in iPTH of greater than or equal to 50%, or either a reduction in iPTH to less than 300 pg/mL or a reduction in iPTH of greater than or equal to 50%.
Time Frame: 24 weeks
Population: The analysis was per protocol. The per-protocol population was defined as all participants who fulfilled inclusion criteria, had intact parathyroid hormone (iPTH) values greater than or equal to 300 pg/mL at baseline, and completed the study with a final iPTH determination. The per-protocol population included 121 participants.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Per-Protocol Population: The per-protocol population was defined as all participants who fulfilled inclusion criteria, had intact parathyroid hormone (iPTH) values greater than or equal to 300 pg/mL at baseline, and completed the study with a final iPTH determination. For this outcome measure, the group evaluated included both participants on hemodialysis receiving paricalcitol injection and those on peritoneal dialysis receiving paricalcitol capsules.
Arm/Group | Per-Protocol Population
Number analyzed (Participants) | 121
days
  Time to achieve iPTH less than 300 pg/mL | 43.80 (41.43)
  Time to achieve 50% or greater reduction in iPTH | 48.68 (43.30)
  Time to achieve either | 40.29 (38.13)

5. Secondary Outcome: Duration of Response to Treatment
Description: Time in days between 2 consecutive visits with a reduction in intact parathyroid hormone (iPTH) of greater than or equal to 50% from the baseline visit.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Per-Protocol Population
Number analyzed (Participants) | 121
days | 65.86 (51.39)

6. Secondary Outcome: Health-related Quality of Life With Paricalcitol Injection or Oral Treatment
Description: Analysis of the differences before and after 24 weeks of treatment in various quality of life measurements for participants on hemodialysis receiving paricalcitol injection and participants on peritoneal dialysis receiving paricalcitol capsules.
Time Frame: Baseline and 24 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules
Number analyzed (Participants) | 32 | 89
Participants
  Mobility-Baseline Score 1 | 13 | 38
  Mobility-Baseline Score 2 | 19 | 47
  Mobility-Baseline Score 3 | 0 | 2
  Mobility-Final Score 1 | 23 | 74
  Mobility-Final Score 2 | 7 | 14
  Mobility-Final Score 3 | 0 | 0
  Personal Care-Baseline Score 1 | 21 | 64
  Personal Care-Baseline Score 2 | 11 | 21
  Personal Care-Baseline Score 3 | 0 | 2
  Personal Care-Final Score 1 | 26 | 79
  Personal Care-Final Score 2 | 4 | 9
  Personal Care-Final Score 3 | 0 | 0
  Daily Activities-Baseline Score 1 | 17 | 35
  Daily Activities-Baseline Score 2 | 15 | 50
  Daily Activities-Baseline Score 3 | 0 | 3
  Daily Activities-Final Score 1 | 26 | 71
  Daily Activities-Final Score 2 | 4 | 16
  Daily Activities-Final Score 3 | 0 | 1
  Pain/Discomfort-Baseline Score 1 | 7 | 24
  Pain/Discomfort-Baseline Score 2 | 24 | 55
  Pain/Discomfort-Baseline Score 3 | 1 | 8
  Pain/Discomfort-Final Score 1 | 25 | 73
  Pain/Discomfort-Final Score 2 | 5 | 15
  Pain/Discomfort-Final Score 3 | 0 | 0
  Anxiety/Depression-Baseline Score 1 | 25 | 34
  Anxiety/Depression-Baseline Score 2 | 7 | 48
  Anxiety/Depression-Baseline Score 3 | 0 | 6
  Anxiety/Depression-Final Score 1 | 26 | 73
  Anxiety/Depression-Final Score 2 | 4 | 15
  Anxiety/Depression-Final Score 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose of study drug through 30 days after the last dose of study drug.
Arm/Group | Paricalcitol Injection | Paricalcitol Capsules
Serious Adverse Events (participants affected / at risk) | 8/38 | 9/109
Other Adverse Events (participants affected / at risk) | 25/38 | 84/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Injection (N=38) | Paricalcitol Capsules (N=109)
Hernia (Gastrointestinal disorders) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Indwelling catheter management (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Injection (N=38) | Paricalcitol Capsules (N=109)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 13 | 31
Hypoparathyroidism (Endocrine disorders) | 10 | 35
Hypothyroidism (Endocrine disorders) | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 3
Vision blurred (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Gingivitis (Gastrointestinal disorders) | 3 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 1
Headache (General disorders) | 6 | 1
Hepatitis (Hepatobiliary disorders) | 5 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Ear infection (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 5
Peritonitis (Infections and infestations) | 0 | 3
Herpes zoster (Infections and infestations) | 1 | 0
Unevaluable event (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Phlebitis (Injury, poisoning and procedural complications) | 7 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 8 | 37
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 24 | 69
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 10
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Oedema (Metabolism and nutrition disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Indwelling catheter management (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 4 | 7
Hypotension (Vascular disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.